CLINICAL TRIAL: NCT02685644
Title: Effects of Laparoscopic Endometrioma Removal on Anti-mullerian Hormone Levels
Brief Title: Association Between Laparoscopic Removal of Endometriomas and Anti-mullerian Hormone Levels
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Erkan Kalafat, Research Assistant, Ankara University
Other Study IDs: 07
Record Dates: First submitted 2016-02-15; First posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Endometriosis; Ovarian Reserve
Keywords: endometrioma; laparoscopy; anti-mullerian hormone; ovarian reserve
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Laparoscopic removal: Patients with endometrioma who will undergo laparoscopic removal of cysts.
  Interventions: Procedure: Laparoscopic removal of cysts

INTERVENTIONS:
Procedure: Laparoscopic removal of cysts — Women with endometrioma lesions will undergo laparoscopic removal. Cysts will be enucleated with blunt dissection of the cyst capsule and following traction, counter traction maneuver. Bipolar coagulation will be used sparsely and suturing will be the predominant choice for achieving bleeding control.

SUMMARY:
Laparoscopic excision of endometriotic cysts is the main stream surgical intervention for treatment of endometriosis. However there is evidence that intervention may effect ovarian reserve by destruction of healthy ovarian tissue during surgery. Available evidence on the topic are contradictory and employed research methodology are diverse. There is need for an adequately powered research with proper methodology to assess actual effects of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women with endometrioma cyst(s)
* Women of age under 35 years old
* Women without any previous ovarian surgery

Exclusion Criteria:

* Combined oral contraceptive or long term GnRH (gonadotropin-releasing hormone) analog use in the preceding 3 months to enrolment
* Having another cystic lesion besides endometrioma
* Need for extensive bipolar coagulation during surgery
* Any anatomical problem preventing evaluation of ovaries with high-resolution ultrasound
* Postoperative pathology excluding endometrioma

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will recruit healthy women besides having endometrioma cysts who will undergo laparoscopic removal of such lesions.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Anti-Mullerian hormone levels | 1 year
  AMH (anti-mullerian hormone) levels will be measured before surgery and during various time points up to 1 year after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Erkan Kalafat, Principal Investigator — Ankara University

IPD SHARING:
Plan to Share IPD: Yes